CLINICAL TRIAL: NCT03724695
Title: Advanced Heart Care at Home (AHCAH); a Pragmatic Randomized Trial for Clinicians Nudged to AHCAH, a Heart Failure Specific Home Palliative Care Services
Brief Title: Advanced Heart Care at Home
Acronym: AHCAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Penn Medicine Center for Health Care Innovation (Unknown); Independence Blue Cross (Other)
Responsible Party: Principal Investigator, Scott Halpern, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 831733
Record Dates: First submitted 2018-10-28; First posted 2018-10-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Palliative Care; Heart Failure; Health Care Utilization; Quality Improvement
MeSH Terms: conditions — Heart Failure; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual Care
- AHCAH Nudge (Experimental): The investigators have developed methods for sending "nudges" to clinicians via secure text messages to primary teams to alert them that their patient was identified as high-risk for 6-month mortality and that an AHCAH liaison would visit their patient to discuss the AHCAH program and to facilitate enrollment if the patient was amenable. The investigators propose that these secure text messages would be sent to the teams of patients randomized to the intervention by the AHCAH liaison within 72 hours of eligibility identification (to allow for the liaison not being available over the weekend). The investigator team will track all aspects of messaging and timing. Clinicians can choose to opt out a patient from the liaison visit and AHCAH enrollment within a two-hour timeframe.
  Interventions: Other: Clinician nudge or opt out approach for AHCAH liaison visit

INTERVENTIONS:
Other: Clinician nudge or opt out approach for AHCAH liaison visit — This study is a "nudge" or opt-out approach of an AHCAH liaison visit to eligible seriously ill HF patients prior to hospital discharge to discuss the AHCAH program and to subsequently facilitate enrolling them in the AHCAH program if they are amenable, compared to the opt-in approach (usual care).
  Arms: AHCAH Nudge

SUMMARY:
End-of-life (EOL) care for heart failure (HF) patients includes high healthcare utilization and costs, in part due to the lack of integration of optimal HF management and home-based palliative care. In a pilot quality improvement project of clinician "nudges" to enroll seriously ill HF patients in a home-based, integrated HF and palliative care platform, the investigators demonstrated decreased healthcare utilization and costs and increased hospice utilization among seriously ill HF patients. The investigators propose a pragmatic randomized trial for clinicians of seriously ill HF patients admitted to three University of Pennsylvania Health System Hospitals, randomly assigning an opt-in approach (usual care) versus a "nudge" or opt-out approach of a visit from an Advanced Heart Care at Home (AHCAH) liaison to clinicians of eligible patients to discuss and enroll in the AHCAH program, to rigorously and scientifically evaluate clinical, utilization, and cost outcomes among high-risk HF patients at the EOL, and to promote physician uptake of best practices.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Reside within Caring Way's geographic catchment
3. Heart Failure ICD code from any previous healthcare encounter (inpatient or outpatient) in the 12 months prior to index hospitalization
4. Admitted to a cardiology or hospitalist service
5. Palliative Connect score greater than 0.3
6. Index hospitalization during study period

Exclusion Criteria:

1. Less than 18 years of age
2. Pregnant women
3. Incarcerated patients
4. Homeless patients
5. Reside outside of Caring Way's geographic catchment
6. Patients without an identifiable primary physician for AHCAH staff to communicate with as determined by the AHCAH liaison via EPIC
7. Prior hospitalization during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Acute care days | 6-12 months
  number of hospitalization days in the University of Pennsylvania Health System

SECONDARY OUTCOMES:
Mortality | 6-12 months
  number of patient deaths after enrollment in AHCAH
Hospice enrollment | 6-12 months
  number of patients who transition from AHCAH to hospice
hospice length of service | 6-12 months
  If transitioned to hospice from AHCAH, number of days on hospice
University of Pennsylvania Health System total acute care cost | 6-12 months
  cost of emergency department visit and/or hospitalization within the UPHS Health system
Pennsylvania total acute care cost | 6-12 months
  cost of emergency department visit and/or hospitalization within Pennsylvania
University of Pennsylvania Health System number of intensive care unit days | 6-12 months
  number of days hospitalized in an intensive care unit within UPHS
Pennsylvania number of intensive care unit days | 6-12 months
  number of days hospitalized in an intensive care unit within hospitals in Pennsylvania
University of Pennsylvania Health System emergency department visits | 6-12 months
  number of emergency department visits within UPHS
Pennsylvania emergency department visits | 6-12 months
  number of emergency department visits within hospitals in Pennsylvania
Use of intravenous diuretics at home | 6-12 months
  Prescription and delivery of intravenous diuretics from Penn Home Infusion Therapy Services and administration of intravenous diuretics by AHCAH nurse
new documentation of goals of care | 6-12 months
  Advance Care Planning documentation within electronic medical record

CONTACTS AND LOCATIONS:
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Russo MJ, Gelijns AC, Stevenson LW, Sampat B, Aaronson KD, Renlund DG, Ascheim DD, Hong KN, Oz MC, Moskowitz AJ, Rose EA, Miller LW; REMATCH Investigators. The cost of medical management in advanced heart failure during the final two years of life. J Card Fail. 2008 Oct;14(8):651-8. doi: 10.1016/j.cardfail.2008.06.005. Epub 2008 Jul 21. PMID 18926436
- [Background] Fang J, Mensah GA, Croft JB, Keenan NL. Heart failure-related hospitalization in the U.S., 1979 to 2004. J Am Coll Cardiol. 2008 Aug 5;52(6):428-34. doi: 10.1016/j.jacc.2008.03.061. PMID 18672162
- [Background] Sahlen KG, Boman K, Brannstrom M. A cost-effectiveness study of person-centered integrated heart failure and palliative home care: Based on a randomized controlled trial. Palliat Med. 2016 Mar;30(3):296-302. doi: 10.1177/0269216315618544. Epub 2015 Nov 24. PMID 26603186
- [Background] Murray SA, Boyd K, Kendall M, Worth A, Benton TF, Clausen H. Dying of lung cancer or cardiac failure: prospective qualitative interview study of patients and their carers in the community. BMJ. 2002 Oct 26;325(7370):929. doi: 10.1136/bmj.325.7370.929. PMID 12399341
- [Background] Warraich HJ, Xu H, DeVore AD, Matsouaka R, Heidenreich PA, Bhatt DL, Hernandez AF, Yancy CW, Fonarow GC, Allen LA. Trends in Hospice Discharge and Relative Outcomes Among Medicare Patients in the Get With The Guidelines-Heart Failure Registry. JAMA Cardiol. 2018 Oct 1;3(10):917-926. doi: 10.1001/jamacardio.2018.2678. PMID 30167645
- [Background] Rogers JG, Patel CB, Mentz RJ, Granger BB, Steinhauser KE, Fiuzat M, Adams PA, Speck A, Johnson KS, Krishnamoorthy A, Yang H, Anstrom KJ, Dodson GC, Taylor DH Jr, Kirchner JL, Mark DB, O'Connor CM, Tulsky JA. Palliative Care in Heart Failure: The PAL-HF Randomized, Controlled Clinical Trial. J Am Coll Cardiol. 2017 Jul 18;70(3):331-341. doi: 10.1016/j.jacc.2017.05.030. PMID 28705314
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Goodlin SJ, Kutner JS, Connor SR, Ryndes T, Houser J, Hauptman PJ. Hospice care for heart failure patients. J Pain Symptom Manage. 2005 May;29(5):525-8. doi: 10.1016/j.jpainsymman.2005.03.005. No abstract available. PMID 15904755
- [Background] Halpern SD. Financial incentives for research participation: empirical questions, available answers and the burden of further proof. Am J Med Sci. 2011 Oct;342(4):290-3. doi: 10.1097/MAJ.0b013e3182297925. No abstract available. PMID 21817878
- [Background] Halpern SD. Prospective preference assessment: a method to enhance the ethics and efficiency of randomized controlled trials. Control Clin Trials. 2002 Jun;23(3):274-88. doi: 10.1016/s0197-2456(02)00191-5. PMID 12057879
- [Background] Halpern SD. Evaluating preference effects in partially unblinded, randomized clinical trials. J Clin Epidemiol. 2003 Feb;56(2):109-15. doi: 10.1016/s0895-4356(02)00598-x. PMID 12654404
- [Background] Halpern SD, Karlawish JH, Berlin JA. The continuing unethical conduct of underpowered clinical trials. JAMA. 2002 Jul 17;288(3):358-62. doi: 10.1001/jama.288.3.358. PMID 12117401
- [Background] Halpern SD. Evidence-based equipoise and research responsiveness. Am J Bioeth. 2006 Jul-Aug;6(4):1-4. doi: 10.1080/15265160600843528. No abstract available. PMID 16885091
- [Background] Halpern SD, Randolph AG, Angus DC. No child left behind: Enrolling children and adults simultaneously in critical care randomized trials. Crit Care Med. 2009 Sep;37(9):2638-41. doi: 10.1097/CCM.0b013e3181a59357. PMID 19602971
- [Background] Kitamura T, Ohtani M, Ueno A, Niijima T. [Biochemical changes after parathyroidectomy in primary hyperparathyroidism. I. Serial changes of Ca, Mg,P, immunoreactive PTH and nephrogenous c-AMP during 2 weeks after parathyroidectomy (author's transl)]. Nihon Hinyokika Gakkai Zasshi. 1981 Feb;72(2):151-8. No abstract available. Japanese. PMID 6265677
- [Background] Halpern SD, Karlawish JH, Casarett D, Berlin JA, Townsend RR, Asch DA. Hypertensive patients' willingness to participate in placebo-controlled trials: implications for recruitment efficiency. Am Heart J. 2003 Dec;146(6):985-92. doi: 10.1016/S0002-8703(03)00507-6. PMID 14660989
- [Background] Halpern SD, Metzger DS, Berlin JA, Ubel PA. Who will enroll? Predicting participation in a phase II AIDS vaccine trial. J Acquir Immune Defic Syndr. 2001 Jul 1;27(3):281-8. doi: 10.1097/00126334-200107010-00011. PMID 11464149
- [Background] Halpern SD, Doyle R, Kawut SM. The ethics of randomized clinical trials in pulmonary arterial hypertension. Proc Am Thorac Soc. 2008 Jul 15;5(5):631-5. doi: 10.1513/pats.200802-019SK. PMID 18625756
- [Background] Rey MM, Ware LB, Matthay MA, Bernard GR, McGuire AL, Caplan AL, Halpern SD. Informed consent in research to improve the number and quality of deceased donor organs. Crit Care Med. 2011 Feb;39(2):280-3. doi: 10.1097/CCM.0b013e3181feeb04. PMID 20975549
- [Background] Carroll R, Antigua J, Taichman D, Palevsky H, Forfia P, Kawut S, Halpern SD. Motivations of patients with pulmonary arterial hypertension to participate in randomized clinical trials. Clin Trials. 2012 Jun;9(3):348-57. doi: 10.1177/1740774512438981. Epub 2012 Mar 2. PMID 22388077
- [Background] Halpern SD, Karlawish JH, Casarett D, Berlin JA, Asch DA. Empirical assessment of whether moderate payments are undue or unjust inducements for participation in clinical trials. Arch Intern Med. 2004 Apr 12;164(7):801-3. doi: 10.1001/archinte.164.7.801. PMID 15078651
- [Background] Faden RR, Kass NE, Goodman SN, Pronovost P, Tunis S, Beauchamp TL. An ethics framework for a learning health care system: a departure from traditional research ethics and clinical ethics. Hastings Cent Rep. 2013 Jan-Feb;Spec No:S16-27. doi: 10.1002/hast.134. No abstract available. PMID 23315888
- [Background] Kerlin MP, Small DS, Cooney E, Fuchs BD, Bellini LM, Mikkelsen ME, Schweickert WD, Bakhru RN, Gabler NB, Harhay MO, Hansen-Flaschen J, Halpern SD. A randomized trial of nighttime physician staffing in an intensive care unit. N Engl J Med. 2013 Jun 6;368(23):2201-9. doi: 10.1056/NEJMoa1302854. Epub 2013 May 20. PMID 23688301
- [Background] Courtright KR, Madden V, Gabler NB, Cooney E, Small DS, Troxel A, Casarett D, Ersek M, Cassel JB, Nicholas LH, Escobar G, Hill SH, O'Brien D, Vogel M, Halpern SD. Rationale and Design of the Randomized Evaluation of Default Access to Palliative Services (REDAPS) Trial. Ann Am Thorac Soc. 2016 Sep;13(9):1629-39. doi: 10.1513/AnnalsATS.201604-308OT. PMID 27348271
- [Background] Department of Homeland Security; Department of Agriculture; Department of Energy; National Aeronautics and Space Administration; Department of Commerce; Social Security Administration; Agency for International Development; Department of Housing and Urban Development; Department of Labor; Department of Defense; Department of Education; Department of Veterans Affairs; Environmental Protection Agency; Department of Health and Human Services; National Science Foundation; Department of Transportation. Federal Policy for the Protection of Human Subjects. Final rule. Fed Regist. 2017 Jan 19;82(12):7149-274. PMID 28106360
- [Background] Kane RL, Finch M, Chen Q, Blewett L, Burns R, Moskowitz M. Post-hospital home health care for Medicare patients. Health Care Financ Rev. 1994 Fall;16(1):131-53. PMID 10140151
- [Background] Stewart S, Marley JE, Horowitz JD. Effects of a multidisciplinary, home-based intervention on unplanned readmissions and survival among patients with chronic congestive heart failure: a randomised controlled study. Lancet. 1999 Sep 25;354(9184):1077-83. doi: 10.1016/s0140-6736(99)03428-5. PMID 10509499
- [Background] Naylor MD, Brooten D, Campbell R, Jacobsen BS, Mezey MD, Pauly MV, Schwartz JS. Comprehensive discharge planning and home follow-up of hospitalized elders: a randomized clinical trial. JAMA. 1999 Feb 17;281(7):613-20. doi: 10.1001/jama.281.7.613. PMID 10029122
- [Result] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885